CLINICAL TRIAL: NCT01579331
Title: Study of Test-retest Reliability of Dynamic Contour Tonometry and Its Correlation With Goldmann Applanation Tonometry
Brief Title: Reliability of Dynamic Contour Tonometry (DCT)
Acronym: DCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luigi Varano, MD - Principal Investigator, M. D., University of Catanzaro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCT01
Record Dates: First submitted 2012-04-15; First posted 2012-04-17 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Intraocular Pressure; Central Corneal Thickness
Keywords: IOP; Tonometry; Pascal; Goldmann; DCT; Dynamic Contour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dynamic Contour Tonometry (Experimental): All recruited volunteers in present study, that underwent diurnal GAT tonometry (3 measures) and 5 DCT measurements.
  Interventions: Device: DCT (PASCAL© Tonometer) IOP and OPA measurement

INTERVENTIONS:
Device: DCT (PASCAL© Tonometer) IOP and OPA measurement — Healthy volunteers recruited among subject that underwent a routine ophthalmologic evaluation or among both students and workers at our clinic, will undergo a series of 5 Dynamic contour tonometries to evaluate eventual differences among measurements.
  Patients will be controlled for 30 days. A diurnal IOP curve performed though GAT, composed of 3 measurements (9am, noon, 4pm) will be taken 1 to 7 days before the DCT. At the end of the DCT measurements a last GAT will be taken to control eventual IOP changes versus previous GAT values obtained through the diurnal curve.
  Other Names: Goldmann Applanation Tonometry (AT900© - Haag-Streit AG, Koeniz, Switzerland); Dynamic Contour Tonometry (PASCAL© Tonometer - Ziemer Ophthalmic Systems AG, Port, Switzerland); Ultrasound pachymeter (Pacline© - Optikon ind., Rome, Italy).

SUMMARY:
Study wants to test reliability Dynamic Contour Tonometry (DCT) in measuring intraocular pressure (IOP) and Ocular Pulse Amplitude (OPA). IOP values obtained with DCT will then be compared with IOP values obtained with Goldmann Applanation Tonometry (GAT), actually the gold standard technique.

DETAILED DESCRIPTION:
Healthy volunteers recruited among subjects who underwent a routine ophthalmologic evaluation or among students and workers both at our clinic, will undergo a series of 5 DCT to evaluate eventual differences among the measurements.

A diurnal IOP curve performed though GAT, composed of 3 measurements (9am, noon, 4pm) will be taken 1 to 7 days before the DCT.

At the end of the DCT measurements a last GAT will be taken to control eventual IOP changes versus previous GAT values obtained through the diurnal curve.

After 3 weeks observers will contact patients to record eventual adverse events. If examiners consider it as necessary, a safety ophthalmological evaluation will then be performed.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects giving a valid consent to be included in this experimentation
* age between 18 and 80 years
* best corrected visual acuity (BCVA) of at least 20/100
* refraction ranging from -6 to +6 dioptres, with an astigmatism ranging from -2 to +2 dioptres

Exclusion Criteria:

* History of refractive surgery or any keratoplasty procedure.
* Corneal opacities or diseases making no suitable applanation tonometry.
* Use of contact lenses. History of glaucoma or ocular hypertension.
* History of diabetic retinopathy staged as severe non-proliferative or worse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
IOP expressed in mmHg | measurements will be taken in a single day, in approximately 30 minutes.
  5 consecutive valid DCT measurements will be taken. After test-retest reliability of these DCT measurements will then be calculated (difference expressed in mmHg between 1st and 5th DCT measurements of IOP. Coefficient of Variation will also be calculated).
OPA expressed in mmHg | measurements will be taken in a single day, in approximately 30 minutes.
  5 consecutive valid DCT measurements will be taken. After test-retest reliability of these DCT measurements will then be calculated (difference expressed in mmHg between 1st and 5th DCT measurements of OPA. Coefficient of Variation will also be calculated).

SECONDARY OUTCOMES:
IOP difference (expressed in mmHG) between first GAT and DCT | partecipants will undergo a GAT diurnal tonometric curve (one day duration) and after one to seven days will undergo 5 DCT (approx. duration 30 minutes)
  The diurnal tonometric curve (i.e. IOP at 9am, noon, 4pm) will be measured using GAT.
  After 1 to 7 days, 5 different IOP measurements recorded every 2 minutes (+/- 1) will be measured at 9am (+/- 15 minutes) using DCT. The difference between GAT and DCT values will be calculated.
IOP difference (expressed in mmHG) between DCT and last GAT | partecipants will undergo 5 DCT and after these, to a single GAT measurement(approx. duration 30 minutes)
  5 different IOP measurements recorded every 2 minutes (+/- 1) will be measured at 9am (+/- 15 minutes) using DCT. After 1-2 minutes a single GAT measurement will be recorded. The difference between GAT and DCT values will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Varano, M. D., Principal Investigator — University of Catanzaro
Locations (1):
- University of Catanzaro - Eye Department, Catanzaro, Catanzaro, Italy